CLINICAL TRIAL: NCT07265219
Title: The Effect of the Health Promotion Model-Based PROBTEC Management Program on Problematic Technology Use in Adolescents: A Randomized Controlled Trial
Brief Title: PROBTEC Program to Manage Problematic Technology Use in Adolescents
Acronym: PROBTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, nesrin arslan, PhD. Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/1261
Record Dates: First submitted 2025-11-22; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Health Promotion Model (HPM); Randomized Controlled Trial; Technology Use; Adolescents
Keywords: Health Promotion Model; problematic technology use; physical activity; randomized controlled trial; adolescents
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded to their group assignment. Although the intervention and control conditions differed in content, students were not informed whether their school had been allocated to the experimental arm or the control arm. The program was delivered within the normal school schedule, and activities were presented in a way that did not disclose group status to the adolescents. Researchers responsible for implementing the intervention were aware of the allocation due to the need to conduct the program; however, participants remained unaware of their assignment throughout the study. Outcome assessments were conducted using standardized scales and objective physical activity monitoring to support unbiased data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: PROBTEC Intervention Group (Experimental): Adolescents in the experimental arm received the PROBTEC Management Program, a structured six-week behavioral intervention based on the Health Promotion Model.
  Interventions: Behavioral: PROBTEC Management Program
- Control: Standard School Routine (No Intervention) (No Intervention): Participants in the control arm continued their usual school schedule without receiving any structured health education or physical activity program related to technology use. They did not participate in any component of the PROBTEC intervention. After the study was completed, informational brochures were provided to ensure ethical equivalence.

INTERVENTIONS:
Behavioral: PROBTEC Management Program — Intervention Description (Distinctive Features) - PROBTEC Program
  The PROBTEC Management Program is a multi-component behavioral intervention specifically designed to address problematic technology use among adolescents within a school setting. Unlike standard health education approaches, this program integrates all core constructs of the Health Promotion Model (HPM) and combines them with structured physical activity strategies and a family-engagement framework. Its distinguishing features include:
  Theory-Driven Structure:
  The entire intervention is explicitly grounded in the Health Promotion Model. Each session targets specific HPM constructs such as perceived benefits, perceived barriers, self-efficacy, situational influences, and interpersonal support. This provides a comprehensive theoretical basis that differentiates the program from generic technology reduction or physical activity programs.
  Combined Digital Behavior + Physical Activity Approach:
  Most existing adolescent inte
  Arms: Experimental: PROBTEC Intervention Group

SUMMARY:
Excessive engagement with digital devices among adolescents has become a significant public health concern, contributing to reduced physical activity and associated health risks. This study assessed the impact of the PROBTEC Management Program-an intervention structured around the Health Promotion Model-on technology-related behaviors and activity levels in adolescents. A randomized controlled trial was implemented in 10 public middle schools in Türkiye with a total sample of 200 students aged 14-15 years. Schools were allocated to either the intervention or control condition using cluster randomization. The intervention spanned six weeks and combined health education sessions, guided physical activity practices, and parent-focused components. Measures were obtained at four time points (baseline, 1 week, 3 months, 6 months) using validated questionnaires, pedometer-based step counts, and the International Physical Activity Questionnaire. Data were analyzed using repeated measures statistical techniques and standardized effect size calculations.

Participants receiving the PROBTEC intervention demonstrated notable improvements over time. Compared with controls, the intervention group exhibited reduced indicators of problematic technology engagement and perceived exercise barriers, alongside increases in perceived exercise benefits, physical activity self-efficacy, and total MET scores.

Findings indicate that the PROBTEC Management Program supports positive behavioral changes by reducing unhealthy technology use and encouraging more active lifestyles among adolescents. The sustained effects observed across the 6-month follow-up period suggest that this school-based, theory-driven model may be a practical and scalable strategy for adolescent health promotion

DETAILED DESCRIPTION:
Problematic technology use has increasingly been recognized as a major behavioral health issue among adolescents, contributing to prolonged sedentary behavior, reduced physical activity, and related negative health outcomes. Although many school-based initiatives address lifestyle or digital well-being independently, few interventions incorporate a comprehensive, theory-guided framework. The PROBTEC Management Program was developed to address this gap by integrating principles from the Health Promotion Model (HPM) to promote healthier technology habits and increase physical activity levels among young people.

This randomized controlled trial evaluated the program's effectiveness in a real-world school setting. Ten public middle schools in Türkiye participated in the study, with cluster randomization used to assign schools to either the intervention or control condition. A total of 200 adolescents aged 14-15 years were included. The intervention consisted of a structured six-week curriculum delivered by trained facilitators and included three core components: (1) health education sessions designed to increase awareness of the risks associated with excessive technology use, (2) guided physical activity practices that encouraged students to incorporate movement into their daily routines, and (3) a parental engagement component aimed at strengthening family support for healthy behaviors.

Outcome measurements were collected at four time points: baseline (T0), immediately after the intervention at 1 week (T1), 3 months post-intervention (T2), and 6 months post-intervention (T3). Technology-related behaviors, perceived benefits and barriers to exercise, and physical activity self-efficacy were assessed using validated instruments. Physical activity levels were evaluated using pedometer-based step counts and the International Physical Activity Questionnaire (IPAQ). Repeated measures statistical analyses were used to examine changes over time, and effect sizes were calculated to estimate the magnitude of intervention effects.

Adolescents who participated in the PROBTEC program showed significant positive changes across all primary outcomes when compared with their peers in the control schools. Reductions in technology addiction scores and perceived exercise barriers were accompanied by increases in perceived benefits of physical activity, self-efficacy for being active, and total MET values. These improvements were evident not only immediately after the intervention but were also maintained throughout the 6-month follow-up period, demonstrating the sustained impact of the program.

Overall, this trial provides evidence that a structured, theory-based, and school-centered intervention can effectively support adolescents in managing digital behaviors while simultaneously promoting physical activity. The PROBTEC Management Program offers a feasible, low-cost, and scalable model that can be integrated into broader school health services. Its combined focus on educational, behavioral, and family-based strategies positions it as a promising approach for addressing the intertwined challenges of technology overuse and physical inactivity in youth populations.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14-15 years
* Volunteering to participate in the study
* Reporting more than two hours of daily screen time
* Able to complete assessments at all required time points

Exclusion Criteria:

* Diagnosed mental disabilities
* Diagnosed physical disabilities
* Presence of chronic illnesses
* Any condition that prevents participation in the intervention or assessments

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Problematic Technology Use Score | Day 0, Day 7, Day 90, Day 180.
  Problematic technology use will be assessed using the Technology Addiction Scale, a validated 32-item scale developed for adolescents. The scale uses a 5-point Likert response format and has four subscales: Social Media Addiction, Instant Messaging Addiction, Online Gaming Addiction, and Website Addiction.
  Total scores range from 0 to 120, with higher scores indicating more severe technology addiction.
  Score interpretation:
  0-24: No addiction
  25-48: Low addiction
  49-72: Moderate addiction
  73-96: High addiction
  97-120: Full addiction
  The scale demonstrated good internal reliability (Cronbach's α = .86 in the original study; α = .97 in the present study).

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Arslan,, PhD, Principal Investigator — Karabuk University; aysun Ardic, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Karabuk University, Faculty of Health Sciences, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves minors and includes sensitive behavioral data that cannot be released under institutional and national data protection regulations. Only aggregated results will be made publicly available.